CLINICAL TRIAL: NCT04795739
Title: Evaluation of ESMO Guidelines Applicability and Adherence in Cancer Pain Management in the Specialist Palliative Care Setting: a Multicenter, Perspective, Observational Study
Brief Title: Evaluation of ESMO Guidelines Applicability and Adherence in Cancer Pain Management in the Palliative Care Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Antea Foundation (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Other Study IDs: PAINSTUDY
Record Dates: First submitted 2021-02-17; First posted 2021-03-12 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cancer Pain; Pain; Cancer
Keywords: Palliative care; Pain; Cancer
MeSH Terms: conditions — Cancer Pain; Pain; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Palliative care (PC) is focused on improving the Quality of Life (QoL) of patients living with a life-threatening illness. Each year, an estimated 40 million people need PC management in the world. In the European Union, it is estimated that about 4,5 million of people are in the need of PC every year, with about 40% affected by malignant neoplasia.

Data from a recent systematic review of the literature report that the prevalence of pain is 66% (95% confidence interval 58-75) in cancer patients with advanced stages of the disease. In 52% of cases, pain was moderate or severe in intensity (NRS, Numeric Rating Scale ≥4). Furthermore, in addition to the basic pain, having characteristics of continuity over time even in the presence of fluctuations in intensity, the presence of acute painful episodes must also be considered, which are defined with the term of Breakthrough Cancer Pain, (BTcP), whose prevalence is estimated between 21 and 59%.

The positive impact on the quality of life of cancer patients of adhering to current guidelines has been amply demonstrated. Recently, new guidelines or recommendations produced by scientific societies have published, including the European Association of Palliative Care, the National Comprehensive Cancer Network and the European Society for Medical Oncology (ESMO).

In clinical facilities directly involved in the treatment of pain in cancer patients, implementing the directives set out in the guidelines appears to be a correct objective for the appropriateness of treatments. Nevertheless, there are no studies in Europe that have evaluated the applicability and adherence to guidelines in the treatment of cancer pain in advanced cancer patients. The present study intends to collect detailed information on the characteristics of pain and the treatment in a population of cancer patients cared by a network of specialized palliative care centers in order to assess the applicability and adherence of the latest European guidelines published by ESMO in 2018 for the treatment of pain in the specific area.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* cancer diagnosis;
* patient enrolled within 48h from admission in PC;
* presence of pain with or without analgesic therapy or absence of pain being already on ATC analgesic therapy;
* life expectancy longer than two weeks;
* written patient informed consent.

Exclusion Criteria:

* diagnosis of primary brain tumor or leukemia (acute or chronic);
* clinical conditions that, at Investigator evaluation, prevent the follow up visits;
* absence of pain without analgesic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with pain in palliative care setting.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-04-07 (Estimated); Study Completion 2022-04-07 (Estimated)

PRIMARY OUTCOMES:
Adherence to ESMO (European Society of Medical Oncology) 2018 Guidelines | Day 14 (final visit).
  The assessment of the adherence of pain treatments to the ESMO 2018 guidelines will be carried out assigning to the 52 recommendations a score of 1 if the recommendation has been satisfied on the patient, 0 if it has not been satisfied and missing if the recommendation was not applicable. A total score will then be calculated for each patient, obtained from the sum of the score for each recommendation divided by the number of applicable recommendations. The percentage of adherence to each single recommendation and to the total of recommendations on all patients will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Casale, Principal Investigator — Antea Foundation
Locations (8):
- Italy (8):
  - Hospice Alba Chiara, Lanciano, Chieti
  - Hospice Torrevecchia Teatina, Torrevecchia Teatina, Chieti
  - Hospice "La Torre sul Colle", Spoleto, Perugia
  - Hospice Carlo Chenis, Civitavecchia, Roma
  - Centro Residenziale di Leniterapia "Roberto Ciabatti", Grosseto
  - Antea Foundation, Roma
  - Centro di Cure Palliative "Insieme nella Cura" - Policlinico Universitario - Campus Bio-Medico (Roma), Roma
  - Fondazione FARO, Torino